CLINICAL TRIAL: NCT07236515
Title: Randomized, Sham-Controlled, Multicenter Investigation of the Leia Sensory Prosthesis on Gait and Balance in Peripheral Neuropathy.
Brief Title: Randomized, Sham-Controlled Investigation of the Leia Sensory Prosthesis in Individuals With Peripheral Neuropathy
Acronym: MYN-L001-001
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MYNERVA AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC.01312:1; Unique Device Identifiers (Other: GS1)
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Neuropathy
Keywords: Peripheral neuropathy; Sensory Prosthesis
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, multicenter.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and outcomes assessors are masked to group allocation (active vs. sham).A subset of care providers responsible for device setup and allocation is unblinded due to practical requirements, while other care providers interacting with participants remain blinded whenever feasible. Investigators at the site have access to allocation information if needed for safety or clinical decision-making.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Device (Experimental): Participants use the active wearable device during the study period.
  Interventions: Device: Active wearable device
- Sham Device (Sham Comparator): Participants use a sham version of the wearable device without active functionality.
  Interventions: Device: Sham wearable device

INTERVENTIONS:
Device: Active wearable device — A non-invasive wearable device used to assess balance, gait, and usability in individuals with peripheral neuropathy.
  Arms: Active Device
Device: Sham wearable device — A sham version of the wearable device without active functionality.
  Arms: Sham Device

SUMMARY:
This study will evaluate a wearable device intended to support balance and gait in adults with peripheral neuropathy. Participants will use the device for a defined period, and outcomes related to safety, usability, and functional performance will be assessed.

DETAILED DESCRIPTION:
This clinical investigation will assess a non-invasive wearable device designed to enhance gait and balance in individuals with peripheral neuropathy. The study will evaluate whether the device can improve balance and gait stability during daily activities, and will also examine safety, comfort, and overall user acceptability over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study procedure.

  * Adults ≥18 years.
  * Clinical diagnosis of peripheral neuropathy.
  * Willingness and ability to attend weekly sessions, perform home use, and return for follow-up.

Exclusion Criteria:

* Age < 18 years at the time of consent.
* Active foot ulcer, infection, or severe dermatological condition at electrode contact sites.
* Cognitive impairment that precludes informed consent or device use.
* Implanted electrical devices or pacemakers.
* Pregnancy
* Usage of other medical devices for the relief of neuropathic symptoms during the trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Functional Gait Assessment (FGA) Total Score | 2 months
  Change in Functional Gait Assessment (FGA) total score (0-30 points) from baseline to 2 months. Higher scores indicate better gait and balance performance.

REFERENCES:
- [Background] Gozzi N, Chee L, Odermatt I, Kikkert S, Preatoni G, Valle G, Pfender N, Beuschlein F, Wenderoth N, Zipser C, Raspopovic S. Wearable non-invasive neuroprosthesis for targeted sensory restoration in neuropathy. Nat Commun. 2024 Dec 30;15(1):10840. doi: 10.1038/s41467-024-55152-7. PMID 39738088